CLINICAL TRIAL: NCT00003838
Title: Non-Myeloablative Allogeneic Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation for Hematologic Malignancies in High Risk Patients and in Patients With Debilitating Hematologic Diseases
Brief Title: Specialized Blood Cell Transplants for Cancers of the Blood and Bone Marrow
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 990050; 99-H-0050; NCT00001875 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2022-10-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-04

CONDITIONS: Myeloproliferative Disorders; Acute Myelogenous Leukemia; Chronic Myelogenous Leukemia; Myelodysplastic Syndrome; Acute Lymphoblastic Leukemia
Keywords: Graft vs. Host Disease; Peripheral Blood Stem Cells; Non-Myeloablative Bone Marrow Transplantation; Engraftment; graft versus leukemia
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Graft vs Host Disease | interventions — Transplantation; Methotrexate; Cyclosporine; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Donor (Other): The HLA matched donor will receive granulocyte colony-stimulating factor (G-CSF) with apheresis collections of PBPC on day 5 and day 6 if required. G-CSF will be administered based on body weight for at least 5, and up to 7 days, subcutaneously.
  Interventions: Drug: G-CSF
- Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality (Experimental): Participants at high risk for transplant related complications and mortality will receive a non-myeloablative preparative regimen of cyclophosphamide 60mg/kg/d x 2 days, and fludarabine 25mg/m^2 intravenously daily x 5 days followed by a peripheral blood hematopoietic progenitor cell graft targeted to deliver >5x10^6 CD34+ cells/kg.
  Interventions: Procedure: T-cell replete PBPC allograft; Drug: Methotrexate; Drug: Cyclosporine
- Group B: Stem Cell Transplant in Debilitating Hematologic Diseases (Experimental): Participants with hematologic diseases associated with reasonable longevity, shown to be curable by allogeneic Bone Marrow Transplant (BMT) but where concern for a high procedural mortality with conventional BMT will receive a non-myeloablative preparative regimen of cyclophosphamide 60mg/kg/d x 2 days, and fludarabine 25mg/m^2 intravenously daily x 5 days followed by a peripheral blood hematopoietic progenitor cell graft targeted to deliver >5x10^6 CD34+ cells/kg.
  Interventions: Procedure: T-cell replete PBPC allograft; Drug: Methotrexate; Drug: Cyclosporine

INTERVENTIONS:
Procedure: T-cell replete PBPC allograft — Subjects will receive a non-myeloablative preparative regimen of cyclophosphamide 60mg/kg/d x 2 days, and fludarabine 25mg/m2 intravenously (IV) over 30 minutes daily x 5 days with or without ATG followed by a PBPC graft targeted to deliver >5x10^6 CD34+ cells/kg.
  Other Names: Peripheral blood hematopoietic progenitor cell (PBPC) transplant
  Arms: Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality; Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Drug: Methotrexate — IV MTX on days +1, +3, and +6 will be given
  Other Names: MTX
  Arms: Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality; Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Drug: Cyclosporine — CSA will be given beginning on day -4 for graft versus host disease prophylaxis. Participants with mixed T-cell chimerism on day 30 will begin a CSA taper. Participants with 100% donor T-cell chimerism by day 30 will be tapered off CSA from days 60 through 100 (25% reduction in dose every 10 days-off by day 100). CSA will not be tapered in any subjects with grade > II acute GVHD regardless of chimerism results. In addition, participants with evidence of disease progression without grade > II GVHD will have CSA discontinued regardless of chimerism results.
  Other Names: CSA
  Arms: Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality; Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Drug: G-CSF — G-CSF will be administered based on body weight for at least 5, and up to 7 days, subcutaneously.
  Other Names: granulocyte colony-stimulating factor (G-CSF)
  Arms: Donor

SUMMARY:
The are a variety of cancerous diseases of the blood and bone marrow that can be potentially cured by bone marrow transplantation (BMT). Diseases like leukemia, lymphoma, and multiple myeloma are among the conditions that can be treated with BMT.

Some patients with these diseases can be treated with medical chemotherapy alone. However, patients who relapse following chemotherapy are usually not curable with additional chemotherapy treatments. The only option known to provide a potential cure if this occurs is BMT.

Allogenic transplants are cells collected from relatives of the patient. The transplant requires additional high intensity chemotherapy and radiation in order to destroy cancerous cells. In the process, many normal bone marrow cells are also destroyed. This is the reason for transplanting stem cells. The stem cells help to build new functioning bone marrow, red cells, white cells, and platelets. In addition, the immune cells from the donor are implanted into the recipient s body and help to fight off infection and kill remaining cancerous cells.

Unfortunately, the powerful doses of chemotherapy and radiation therapy associated with allogenic BMT have toxic side effects and often make BMTs too dangerous to attempt in many patients.

In order to reduce the complications of BMT, and make it a safer available option for patients with cancers of the blood and bone marrow, researchers have developed a new approach to the BMT.

In this study researchers plan to use stem cells collected from the blood stream of patient s relatives rather than from the bone marrow (blood progenitor/stem cell transplant). In addition, researchers plan to use low doses of chemotherapy and no radiation therapy to reduce side effects. The majority of the cancer killing effect will be the responsibility of the stem cell transplant rather than the chemotherapy.

DETAILED DESCRIPTION:
Patients with malignant and non-malignant hematologic diseases including severe aplastic anemia (SAA), paroxysmal nocturnal hemoglobinuria (PNH), myelodysplastic syndrome (MDS), acute and chronic leukemias, Hodgkin's and non-Hodgkin's lymphoma and multiple myeloma (MM) can now be cured by allogeneic bone marrow transplantation (BMT). This curative effect has been ascribed to the use of high dose chemo-radiotherapy and the anti-tumor or anti-bone marrow effect of the allograft. Dose intensification of conditioning regimens in attempts to reduce disease recurrence has been largely unsuccessful because of increased toxicity and mortality. Indeed, most evidence now points to donor-derived T-cells as being the principal modality leading to the complete eradication of both malignant and non-malignant host hematopoietic cells.

The assumption that successful allogeneic BMT relies on the myeloablative effect of intensive but hazardous chemo-radiotherapy has largely restricted this therapeutic modality to patients with malignant or life-threatening hematologic disorders under the age of 55 years. Treatment-related mortality increases substantially with age, prior intensive treatment with chemo-radiotherapy, worsening performance status, and co-morbid medical conditions. An unacceptable risk of death from conventional BMT renders many patients ineligible for what may otherwise be curative therapy.

Several in vitro studies have demonstrated the existence of donor-derived CD4 and CD8 positive lymphocytes with specific reactivity for the patient s leukemia. These cells provide a potent graft-versus-leukemia (GVL) effect. This GVL effect is best seen in patients with CML relapsing after BMT, where a single infusion of donor lymphocytes has been shown to induce complete remission. In addition to the potent anti-leukemia effect of these cells, there is now strong evidence that donor T-cells are capable of completely eradicating residual host hematopoietic cells in a non-myeloablative transplant setting (graft-versus-marrow) leading to successful and complete donor hematopoietic engraftment.

Non-myeloablative allogenic peripheral blood stem cell transplants are currently being investigated in phase I/II trials assessing engraftment efficacy and toxicity at a number of transplant centers. Preliminary data, including our own experience with greater than 150 patients undergoing this type of procedure, have shown a high rate of complete donor engraftment with a low toxicity profile. Two recent studies investigating non-myeloablative allo-transplantation in standard risk patients revealed an extremely low rate of transplant-related complications and mortality.

The decreased risk of transplant-related complications associated with non-myeloablative transplants expands the eligibility of transplant candidates as well as opens the possibility to evaluate non-myeloablative regimens in patients at high risk for complications with standard transplantation. Besides hematologic malignancies, allogeneic BMT has been shown to be curative in a number of debilitating hematologic diseases which may behave in a relatively indolent fashion, such as paroxysmal nocturnal hemoglobinuria (PNH) and refractory anemia (RA) or refractory anemia with ringed sideroblasts (RARS). However, the 30% risk of treatment-related mortality (TRM) with standard myeloablative allotransplantation usually precludes these patients from potentially curative therapy, because of concerns about shortening life in patients with these disorders. In this protocol we investigate non-myeloablative allogeneic peripheral blood stem cell (PBSC) transplantation in two groups of subjects where standard allogeneic transplantation is considered to have unacceptable toxicity.

Group A: Subjects with hematologic malignancies with factors putting them at high risk for transplant related complications and mortality, including prior intensive chemo-radiotherapy and co-morbid diseases.

Group B: Subjects with hematologic diseases (both clonal and non-clonal) associated with reasonable longevity not currently considered for allogeneic BMT because of prohibitive procedural mortality with conventional BMT (enrollment closed October 2010).

In this protocol, eligible subjects are treated with an allogeneic PBSC transplant from an HLA identical or single HLA antigen-mismatched family donor, using an intensive immunosuppressive regimen without myeloablation in an attempt to decrease the transplant related toxicities while preserving the anti-malignancy and/or anti-host marrow effect of the graft. The low intensity non-myeloablative conditioning regimen should provide adequate immunosuppression to allow stem cell and lymphocyte engraftment. T-cell replete, donor-derived, granulocyte colony stimulating factor (G-CSF)-mobilized PBSCs will be used to establish hematopoietic and lymphoid reconstitution. We will add back lymphocytes in recipients with less than 100% donor T-cell chimerism in an attempt to prevent graft rejection and enhance a graft-versus-malignancy effect.

The primary endpoint of this study is transplant related mortality (200 day survival). Other end points include engraftment, degree of donor-host chimerism, incidence of acute and chronic graft versus host disease (GVHD), transplant related morbidity as well as disease-free and overall survival.

ELIGIBILITY:
* INCLUSION CRITERIA - Recipients:

Group A: Subjects at high risk for transplant related complications and mortality as defined below:

Ages 10 to 75 (both inclusive) with a history of one of the following:

* Treatment with dose intensive chemotherapy and/or radiotherapy
* Previous history of allo/auto transplant
* History of multiple myeloma or extramedullary plasmacytoma
* Chronic disease or co-morbid medical condition including subjects with symptoms or signs of significant pulmonary disease, hepatic disease, kidney disease, cardiac disease or disease of other organ systems which would result in increased risk of morbidity or death from a standard myeloablative transplant.

Diseases to be included:

* CML chronic phase
* Acute lymphoblastic leukemia (ALL), all subjects in complete or partial remission.
* AML: AML in first complete or partial remission Exceptions: AML with good risk karyotypes: AML M3 t(15:17), AML M4Eo (inv. 16), AML t(8;21). All AML in second or subsequent complete remission.
* MDS: refractory anemia with excess blasts (RAEB), or chronic myelomonocyte leukemia (CMML).
* Myeloproliferative diseases associated with either cytopenia or uncontrolled proliferation.
* CLL or small lymphocytic lymphoma (SLL) with bulky or progressive disease despite prior treatment with chemotherapy which includes purine analogs.
* NHL

A) Intermediate or high grade relapsed or progressive despite treatment with standard therapy ineligible for autologous PBSC transplant.

B) NHL intermediate or high grade relapsing despite prior autologous transplant.

C) Low grade follicular or small lymphocytic lymphoma (1) high risk patients who have relapsed following conventional chemotherapy, (2) relapsed following autologous marrow or PBSC transplant, or (3) chemo resistant disease.

D) Mantle cell lymphoma

E) NHL intermediate or high grade with concurrent BCL2 and MYC translocations who are at high risk for relapsed and who have low survival with conventional chemotherapy.

* HD, relapsed after prior autologous transplant or after 2 or more combination chemotherapy regimens and ineligible for autologous PBSC transplant.
* EBV driven lymphoproliferative disorders progressing despite standard therapies.
* MM: MM subjects must be between the ages of 8 and 65 (both inclusive)
* Mycosis fungoides, which has been shown to be amenable to allogeneic stem cell transplants.

Group B: (Closed to enrollment Oct 2010) Subjects with hematologic diseases associated with reasonable longevity, shown to be curable by allogeneic BMT but where concern for a high procedural mortality with conventional BMT may delay or prevent such treatment.

Ages 8 to 80 (both inclusive) with a history of one of the following

* PNH associated with either life-threatening thrombosis, cytopenia, transfusion dependence or recurrent and debilitating hemolytic crisis.
* Aplastic anemia or PRCA (acquired or congenital) in subjects associated with transfusion dependence and/or neutropenia who are not candidates for or who have failed immunosuppressive therapy
* RA or RARS MDS subjects who have associated transfusion dependence and/or neutropenia.

Ability to comprehend the investigational nature of the study and provide informed consent. The procedure will be explained to subjects age 8-17 years with formal consent being obtained from parents or legal guardian.

Availability of HLA identical or single HLA locus mismatched family donor

INCLUSION CRITERIA - Donor:

HLA identical or single HLA mismatched family donor

Age greater than or equal to 2 up to 80 years old

Weight greater than or equal to 18 kg

Ability of donor or guardian of donor to comprehend the investigational nature of the study and provide informed consent.

EXCLUSION CRITERIA - Recipient - any of the following:

Pregnant or lactating

Group A: age less than 10 or greater than 75 (multiple myeloma age less than 8 or greater than 65);

Group B: Age less than 8 or greater than 80 years.

ECOG performance status of 3 or more (See NIH Bone and Marrow Consortium Supportive Care Guidelines for Allogeneic Hematopoietic Stem Cell Transplant Recipients - http://intranet.cc.nih.gov/bmt/_pdf/ECOG_Karnofsky_Lansky_Scales.pdf)

Psychiatric disorder or mental deficiency severe as to make compliance with the BMT treatment unlikely and making informed consent impossible

Major anticipated illness or organ failure incompatible with survival from PBSC transplant

Diffusion capacity of carbon monoxide (DLCO) less than 40% predicted.

Left ventricular ejection fraction: less than 30%.

Serum creatinine greater than 2.5 mg/dl or creatinine clearance less than 50 cc/min by 24 hr urine collection

Serum bilirubin greater than 4 mg/dl, transaminases greater than 5x upper limit of normal,

Other malignant diseases liable to relapse or progress within 5 years.

EXCLUSION CRITERIA - Donor - any of the following:

Pregnant or lactating

Donor unfit to receive G-CSF and undergo apheresis (uncontrolled hypertension, history of congestive heart failure or unstable angina, thrombocytopenia)

HIV positive donor. Donors who are positive for hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV I/II) will be used at the discretion of the investigator following counseling and approval from the recipient

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 1999-04-15 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Childs, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Buchan A, Merideth MA, Childs RW, Stratton P. Novel management of vaginal chronic graft-versus-host disease causing haematometra and haematocolpos. BMJ Case Rep. 2018 Apr 28;2018:bcr2017222720. doi: 10.1136/bcr-2017-222720. PMID 29705733
- [Derived] Pantin J, Tian X, Shah AA, Kurlander R, Ramos C, Cook L, Khuu H, Stroncek D, Leitman S, Barrett J, Donohue T, Young NS, Geller N, Childs RW. Rapid donor T-cell engraftment increases the risk of chronic graft-versus-host disease following salvage allogeneic peripheral blood hematopoietic cell transplantation for bone marrow failure syndromes. Am J Hematol. 2013 Oct;88(10):874-82. doi: 10.1002/ajh.23526. Epub 2013 Sep 3. PMID 23813900
- [Derived] Sri T, Merideth MA, Pulanic TK, Childs R, Stratton P. Human papillomavirus reactivation following treatment of genital graft-versus-host disease. Transpl Infect Dis. 2013 Aug;15(4):E148-51. doi: 10.1111/tid.12098. Epub 2013 May 28. PMID 23710698
- [Derived] Baskar S, Suschak JM, Samija I, Srinivasan R, Childs RW, Pavletic SZ, Bishop MR, Rader C. A human monoclonal antibody drug and target discovery platform for B-cell chronic lymphocytic leukemia based on allogeneic hematopoietic stem cell transplantation and phage display. Blood. 2009 Nov 12;114(20):4494-502. doi: 10.1182/blood-2009-05-222786. Epub 2009 Aug 10. PMID 19667400
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1999-H-0050.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Donor: The HLA matched donor will receive granulocyte colony-stimulating factor (G-CSF) with apheresis collections of peripheral blood progenitor cells on day 5 and day 6 if required.
  G-CSF will be administered based on body weight for at least 5, and up to 7 days, subcutaneously.
Period: Overall Study
Arm/Group | Donor | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Started | 102 | 43 | 57
Completed | 102 | 18 | 49
Not Completed | 0 | 25 | 8
Not completed — Death | 0 | 12 | 7
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Disease Progression | 0 | 12 | 0

BASELINE CHARACTERISTICS:
Groups:
- Donor: The HLA matched donor will receive granulocyte colony-stimulating factor (G-CSF) with apheresis collections of PBPC on day 5 and day 6 if required.
  G-CSF: G-CSF will be administered based on body weight for at least 5, and up to 7 days, subcutaneously.
- Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality: Participants at high risk for transplant related complications and mortality will receive a non-myeloablative preparative regimen of cyclophosphamide 60mg/kg/d x 2 days, and fludarabine 25mg/m^2 intravenously (IV) daily x 5 days followed by a peripheral blood hematopoietic progenitor cell (PBPC) graft targeted to deliver >5x10^6 CD34+ cells/kg
- Group B: Stem Cell Transplant in Debilitating Hematologic Diseases: Participants with hematologic diseases associated with reasonable longevity, shown to be curable by allogeneic BMT but where concern for a high procedural mortality with conventional Bone Marrow Transplant will receive a non-myeloablative preparative regimen of cyclophosphamide 60mg/kg/d x 2 days, and fludarabine 25mg/m^2 intravenously (IV) daily x 5 days followed by a peripheral blood hematopoietic progenitor cell (PBPC) graft targeted to deliver >5x10^6 CD34+ cells/kg
- Total: Total of all reporting groups
Arm/Group | Donor | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases | Total
Number analyzed (Participants) | 102 | 43 | 57 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 2 | 11 | 26
  Between 18 and 65 years | 87 | 41 | 45 | 173
  >=65 years | 2 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 18 | 22 | 89
  Male | 53 | 25 | 35 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 10 | 25 | 69
  Not Hispanic or Latino | 68 | 30 | 32 | 130
  Unknown or Not Reported | 0 | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 9 | 0 | 9 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 17 | 7 | 9 | 33
  White | 43 | 26 | 14 | 83
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 33 | 8 | 25 | 66
Region of Enrollment [Number; unit: participants]
  United States | 102 | 43 | 57 | 202

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Transplant Related Mortality
Description: Number of Participants who experienced transplant related mortality by Day 200
Time Frame: 200 days
Population: The analyses included only those participants who had a transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Number analyzed (Participants) | 43 | 57
Participants | 5 | 4

2. Secondary Outcome: Number of Participants With Complete Donor Myeloid (CD34+) and T-cell (CD3+) Chimerism
Description: Number of participants with complete donor myeloid chimerism. Myeloid (CD34+) and T-cell (CD3+) chimerisms were determined by PCR analysis of short tandem repeats (STR). Complete donor chimerism is defined as >95% donor-derived cells in the peripheral blood in a specific lineage.
Time Frame: Up to Day 100
Population: Alive participants who had a transplant with data available for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Number analyzed (Participants) | 31 | 57
Participants
  complete donor myeloid (CD34+) chimerism | 29 | 55
  complete T-cell (CD3+) chimerism | 30 | 56

3. Secondary Outcome: Median Days to Neutrophil Engraftment
Description: Median days to neutrophil recovery. Neutrophil recovery is defined as the first day of two consecutive days in which the ANC was 500 K/ml or greater unsupported by growth factors or granulocyte transfusion.
Time Frame: Day 30
Population: Alive participants who had a transplant with data available for analysis
Measure: Median (Full Range); unit: Days
Arm/Group | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Number analyzed (Participants) | 39 | 56
Days | 14 [7 to 22] | 15 [6 to 24]

4. Secondary Outcome: Number of Participants Who Experienced Acute GVHD Grades II-IV
Description: Number of participants who experienced acute GVHD grades II-IV
  Acute-GVHD was graded and staged prospectively using criteria from the 1994 Consensus Conference on Acute-GVHD Grading.
  Grades are defined as:
  Grade II: Skin = rash on 25-50 percent body surface area; Liver = Total Bilirubin 3.1-6.0 mg/dL; Lower GI = Diarrhea 1001-1500 mL/day.
  Grade III: Skin = Rash on >50% of body surface; Liver = Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI = Diarrhea > 1500 mL/day.
  Grade IV: Skin = Generalized erythroderma plus bullous formation; Liver = Total Bilirubin >15 mg/dL; Lower GI = Severe abdominal pain with or without ileus.
  Grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: Up to Day 100
Population: analysis performed as intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Number analyzed (Participants) | 43 | 57
Participants
  Grade II | 6 | 16
  Grade III-IV | 14 | 18

5. Secondary Outcome: Number of Participant Who Experienced Chronic Graft Versus Host Disease Following Stem Cell Transplant
Description: Number of participant who experienced chronic graft versus host disease (GVHD) following stem cell transplant
  The diagnosis of clinical features of chronic-GVHD was determined prospectively and classified retrospectively into limited or extensive based on the Revised Seattle Classification. Chronic GvHD severity categorized as "limited" is defined as: localized skin lesions with or without limited hepatic involvement and "extensive" is defined as: generalized skin involvement, major hepatic complications, or involvement of any other organ.
Time Frame: Day 100 up to 3 years
Population: The analyses included only those participants that engrafted and survived over 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Number analyzed (Participants) | 38 | 55
Participants
  Limited | 12 | 13
  Extensive | 19 | 27

6. Secondary Outcome: Number of Participants Overall Survival
Description: Number of participants overall survival. Overall survival is defined as number participants alive following stem cell transplant
Time Frame: enrollment to date of death, up to 5 years
Population: The analyses included only those participants that had a stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Number analyzed (Participants) | 43 | 57
Participants | 17 | 48

7. Secondary Outcome: Number of Participants That Remained Disease-free Survival
Description: Number of participants that remained Disease-free survival following stem cell transplant. Disease-free survival is defined as survival free of disease relapse or disease progression following stem cell transplant.
Time Frame: Up to 5 years
Population: The analyses included only those participants that had a stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases
Number analyzed (Participants) | 43 | 57
Participants | 26 | 56

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases | Donor
All-Cause Mortality (participants affected / at risk) | 26/43 | 9/57 | 0/101
Serious Adverse Events (participants affected / at risk) | 41/43 | 47/57 | 1/101
Other Adverse Events (participants affected / at risk) | 0/43 | 0/57 | 0/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Group A: Stem Cell Transplant in High Risk for Transplant Related Complications and Mortality (N=43) | Group B: Stem Cell Transplant in Debilitating Hematologic Diseases (N=57) | Donor (N=101)
Acute Gastrointestional Graft Verses Host Disease (Immune system disorders) | 8 (8) | 9 (14) | 0/0 (0)
Acute Graft verses Host Disease of Skin (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Acute on Chronic Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute right parietal/occipital lobe hemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Acute Upper Gastrointestional Graft Verses Host Disease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Adenoviral enteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Allergic reaction to medication (General disorders) | 1 (1) | 0 (0) | 0 (0)
Alveolar infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Appendecitis (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aspergillosis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
ATG induced anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
ATG induced reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Axonal polyneuropathy cyclosporine induced (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 7 (8) | 9 (18) | 0 (0)
Bilateral Lung Infiltrates (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bone Marrow positive for megakaryocytes (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter Related Thrombosus (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic Graft Verses Host Disease (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Graft Verses Host Disease of Liver (Immune system disorders) | 2 (2) | 1 (1) | 0 (0)
Chronic Graft Verses Host Disease of Lungs (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic Graft Verses Host Disease of Skin (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic left ankle ulcer osteomyelitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Clostridioides difficile (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
CMV colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
CMV Reactivation (Infections and infestations) | 3 (3) | 4 (4) | 0 (0)
Cold Symptoms (Investigations) | 1 (1) | 0 (0) | 0 (0)
Community Acquired Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dacryocystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Diffuse Alveolar hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Disease progression (General disorders) | 3 (3) | 0 (0) | 0 (0)
Disseminated zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Emesis (General disorders) | 1 (1) | 1 (1) | 1 (1)
Engraftment Syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Enterovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erosive gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Exacerbation of Chronic Obstructive Pulmonary Disease with Upper Respirtory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 4 (4) | 4 (4) | 0 (0)
Fluid Overload (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Glomerular microangiopathic thrombosis suggestive of hemolytic uremia syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Graft verses host disease reactivation (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Hemoptysis (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster reactivation (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Hyperglycemia (Investigations) | 1 (1) | 4 (4) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Idiopathic Terminal Ileitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Increased Liver Function Tests (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Ingrown toe nail positive for Staphylococcus aureus and beta-hemolytic Strep A (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Interstitial Pneumonitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Intracranial bleed (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Klebsiella Pneumonia in Urine (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Left Limb Ischemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lesion on lip positive for septate hyphae and dichotomous branching (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Line Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Loss of balance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lower Extremity Edema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Mallory Weiss tear (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mucoepidermoid carcinoma of hard pallate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mucomucosis of lungs (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (General disorders) | 1 (1) | 0 (0) | 1 (1)
Necrotizing fasciitis by Clostridium septicum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neutropenic fever (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Occipital hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Odynophagiam skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Oral Graft verses Host Disease (Immune system disorders) | 2 (2) | 0 (0) | 0 (0)
Oral Herpes simplex virus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 5 (5) | 1 (2) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Parainfluenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pericardectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (12) | 7 (8) | 0 (0)
Pneumonmediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Positive for Hookworm egg (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Positive Pseudomonas Aeruginosa Blood Cultures (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PRES (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Refractory Graft verses host disease (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Rhinovirus (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Rigors (General disorders) | 1 (1) | 0 (0) | 0 (0)
Salmonella Food Poisoning (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 3 (4) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 5 (6) | 0 (0)
Skin Abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Small bowell obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Steriod Refractory Gastrointestional Graft verses host disease (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Subdural hematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0)
Thrombocytopenia with giant platelets (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tooth pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Toxoplasmosis gondii of the right eye (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Transient Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Transjugular Biopsy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper Respirtory Infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 2 (3) | 0 (0)
Viral gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection on wrist (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Group B: Stem Cell Transplant in Debilitating Hematologic Diseases was closed to enrollment in 2010.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT00003838/Prot_SAP_001.pdf